CLINICAL TRIAL: NCT05813964
Title: A Randomized Controlled Trial to Evaluate the Efficacy, Acceptability and Safety of Event-driven Pre-exposure Prophylaxis for HIV Using TAF/FTC in Men Who Have Sex With Men in Thailand and France
Brief Title: Efficacy, Acceptability and Safety of Event-driven HIV PrEP Using TAF/FTC in MSM in Thailand and France.
Acronym: SimpPrEP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Chiang Mai University, Thailand (Unknown); Ministry of Health, Thailand (Other Government); Assistance Publique - Hôpitaux de Paris, FRANCE (Unknown); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 0029s; 2022-502931-20 (EudraCT Number)
Record Dates: First submitted 2023-03-02; First posted 2023-04-14 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: HIV/AIDS
Keywords: PrEP exposure prophylaxis (PrEP); On-demand; Event-driven; TAF
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: This is a phase III, international, multicenter, open-label, parallel-group, randomized, controlled trial among cis men who have sex with men.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Event-driven PrEP with TDF/FTC (Active Comparator): Participants randomly assigned to the event-driven TDF/FTC arm will be instructed to take a loading dose of two single tablets containing coformulated TDF/FTC (300/200mg) 2 to 24 hours before sexual intercourse, followed by a third pill 24 hours after the first drug intake and a fourth pill 24 hours later. In case of daily sexual intercourses, they will be instructed to take one pill per day until the last sexual intercourse, then to take the two post-exposure pills.
  Interventions: Drug: TDF/FTC 300mg/200mg fixed-dose combination tablets
- Event-driven PrEP with TAF/FTC (Experimental): Participants randomly assigned to the event-driven TAF/FTC arm will be instructed to take one single tablet containing coformulated TAF/FTC (25/200mg) with or without food 2 to 24 hours before sexual intercourse followed by a second pill 24 hours after the first drug intake. In case of daily sexual intercourses, they will be instructed to take one pill per day until the last sexual intercourse and then a last pill 24 hours later.
  Interventions: Drug: TAF/FTC 25mg/200mg fixed-dose combination tablets

INTERVENTIONS:
Drug: TDF/FTC 300mg/200mg fixed-dose combination tablets — Event-driven dosing regimen
  Other Names: Truvada
  Arms: Event-driven PrEP with TDF/FTC
Drug: TAF/FTC 25mg/200mg fixed-dose combination tablets — Event-driven dosing regimen.
  Other Names: Descovy
  Arms: Event-driven PrEP with TAF/FTC

SUMMARY:
The purpose of this study is to evaluate the efficacy, acceptability, and safety of a simplified event-driven pre-exposure prophylaxis of HIV based on oral TAF/FTC in HIV-uninfected cisgender men who have sex with men (MSM).

Primary objective: To assess the efficacy of emtricitabine 200 mg + tenofovir alafenamide 25 mg (F/TAF), taken 2 to 24 hours before sexual intercourse followed by a second dose 24 hours after the first intake, in reducing the risk of HIV acquisition in MSM relative to the background HIV incidence rate.

DETAILED DESCRIPTION:
The study will enroll HIV-uninfected MSM at risk for acquiring HIV infection. Participants will be enrolled over 2 years and followed up until the closure of the clinical study. Therefore, the follow up duration will be up to 3 years for first enrollees and up to1 year for the last enrollee. The study will be implemented in Thailand (60% of participants) and France (40%).

Participants will be randomly assigned to one of two regimens:

* Experimental Arm (F/TAF): one tablet of the fixed-dose combination of emtricitabine (FTC) 200 mg + tenofovir alafenamide (TAF) 25mg, 2 to 24 hours before sexual intercourse followed by a second tablet 24 hours after the first intake.
* Control Arm (F/TDF): two tablets of the fixed-dose combination of emtricitabine (FTC) 200 mg + tenofovir disoproxil fumarate (TDF) 300 mg, 2 to 24 hours before sexual intercourse followed by a third tablet 24 hours after the first drug intake and a fourth tablet 24 hours later.

Participants will attend up to 15 study visits throughout the study. Visits may include physical examinations, blood collection, urine collection, and swabs collection (oral and rectal). At the end of their study participation, all participants will be transitioned to locally available HIV prevention services, including PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Male at birth age ≥ 18 years old
* Reporting having sex with men
* Negative 4th generation HIV-1 and HIV-2 test
* Reporting condomless anal sex with men not more often than two days during the previous month and able to plan their sexual activity
* Risk of HIV acquisition based on self-report of at least one of the following behaviors during the 6 months before enrollment: condomless anal sex with at least 2 different sexual partners, sexually transmitted infection (rectal chlamydia and/or rectal gonorrhea and/or syphilis), provided or received money goods or favor in exchange of sex, binge drinking or use of non-injectable recreational drugs.
* Consenting to participate and agreeing to follow the clinical trial procedures, including adherence to study visits every 3 months
* In France: Person affiliated with or benefiting from a social security system (article L1121-11of the public health code in France)

Non-inclusion criteria:

* Symptoms and/or clinical signs consistent with an acute HIV infection
* Women and trans women
* Taking feminizing hormone therapy
* Positive HIV test result at screening or enrollment even if HIV infection is not confirmed
* Positive hepatitis B surface antigen test
* ALT or AST > 4 ULN
* Estimated glomerular filtration rate < 60mL/min/1.73m²
* History of chronic kidney disease, osteoporosis, osteopenia or pathological fracture not related to trauma
* Hypersensitivity to the study products F/TDF or F/TAF
* Past or concurrent participation in a HIV vaccine trial or concurrent participation in another clinical trial without the agreement of the principal investigators of the two trials
* Use of intravenous drugs within the last 12 months
* Person under legal guardianship
* Not likely to comply with the clinical trial procedures or with any condition incompatible with study participation, upon the investigator's judgement.
* Ongoing Post-Exposure Prophylaxis (PEP) for HIV

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men
Enrollment: 524 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of F/TAF | All along the study
  Number of HIV infections defined by the presence of HIV ribonucleic acid (RNA) in plasma through study completion (an average of two years) in the event-driven F/TAF arm.

SECONDARY OUTCOMES:
Efficacy of F/TDF | All along the study
  Number of HIV infections defined by the presence of HIV ribonucleic acid (RNA) in plasma through study completion (an average of two years) in the event-driven F/TDF arm.
Acceptability of F/TAF versus F/TDF | At 1 and at 2 years of follow up.
  Satisfaction score assessed by a self-administrated study medication satisfaction questionnaire.
Safety of F/TAF versus F/TDF | All along the study
  1. Numbers of participants experiencing, through study completion (an average of 2 years):
     * at least one Grade 3 or 4 treatment-related adverse event as graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events [Corrected Version 2.1 July 2017],
     * at least one serious adverse event as graded using the same tables.
  2. Change from baseline in estimated glomerular filtration rate at 1, 2, and 3 years.
  3. Change from baseline in body weight at 1, 2, and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffroy LIEGEON, Study Director — Infectious Diseases Department, Saint-Louis Hospital, Paris, France; Sumet ONGWANDEE, Study Director — Office of the Senior Expert Committee, Department of Disease Control, Ministry of Public Health, Nonthaburi, Thailand
Locations (4):
- France (2):
  - AP-HP - Hospital Lariboisière, Paris
  - AP-HP - Hôpital Saint-Louis, Paris
- Thailand (2):
  - MPlus Clinic, Chiang Mai
  - STIs Clinic of the Office of Disease Prevention and Control Region 1, Chiang Mai

IPD SHARING:
Plan to Share IPD: No